CLINICAL TRIAL: NCT06719947
Title: High-Definition Transcranial Direct Current Stimulation (HD-tDCS) in Amyotrophic Lateral Sclerosis: A Multicenter Randomized Controlled Trial
Brief Title: HD-tDCS in Amyotrophic Lateral Sclerosis: A Multicenter Randomized Controlled Trial
Acronym: tDCS-ALS
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Guilherme Augusto de Freitas Fregonezi, Professor, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD-tDCSALS; U1111-1306-808 (Other: Universal Test Number (UTN))
Record Dates: First submitted 2024-11-30; First posted 2024-12-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis (ALS); Central Nervous System Diseases; Electric Stimulation Therapy; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HD-tDCS Group (Experimental): Patients randomly included in this group will receive 10 sessions of anodal HD-tDCS stimulation. The intervention will take place at the participant's home, with electrodes positioned in a circular arrangement-one central electrode and four peripheral electrodes-over the cortical representation zone of the left primary diaphragmatic motor cortex, with a continuous current applied
  Interventions: Device: Active HD-tDCS
- HD-tDCS sham group (Placebo Comparator): Patients randomly included in this group will receive 10 sessions of sham HD-tDCS stimulation. The intervention will take place at the participant's home, with electrodes positioned in a circular arrangement-one central electrode and four peripheral electrodes-over the cortical representation zone of the left primary diaphragmatic motor cortex. Only an initial 30-second ramp stimulus will be applied, followed by a non-effective current
  Interventions: Device: Simulated HD-tDCS

INTERVENTIONS:
Device: Active HD-tDCS — 10 sessions of anodal HD-tDCS stimulation (neurostimulator coupled with a 4x1 HD-tDCS multichannel adapter) with a defined electrical current intensity over the cortical representation zone of the left diaphragmatic motor cortex
  Arms: Active HD-tDCS Group
Device: Simulated HD-tDCS — 10 sessions of sham anodal HD-tDCS stimulation (neurostimulator coupled with a 4x1 HD-tDCS multichannel adapter) over the cortical representation zone of the left diaphragmatic motor cortex. The device will provide a 30-second ramp and then maintain a minimal, non-effective continuous current
  Arms: HD-tDCS sham group

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a nervous system disease that causes muscle weakness and rapidly progresses to the loss of mobility and functionality. Studies suggest that High-Definition Transcranial Direct Current Stimulation (HD-tDCS) is a technique for modulating motor cortical hyperexcitability. However, evidence on the use of HD-tDCS as a neuromodulator of the diaphragmatic motor cortex in people with ALS is inconclusive.

DETAILED DESCRIPTION:
A multicenter, randomized controlled clinical trial will be conducted. Participants will be randomized into two groups: the HD-tDCS group (gTDCS) and the sham tDCS group (gSham). The intervention protocol will assess the effects of HD-tDCS on respiratory parameters and ALS progression. The study will include individuals of both sexes, aged 18 to 80 years, with a clinical diagnosis of ALS, evaluated before, during, and after the home-based HD-tDCS protocol. The electrodes will be positioned in a circular arrangement over the primary diaphragmatic motor cortex, applying a continuous anodal current intensity. For placebo comparison, only an initial 30-second ramp stimulus will be applied, followed by a minimal current, resulting in no significant intervention. The intervention will be conducted at the participant's home, once daily, five days per week, for two weeks. Patients will undergo evaluations of lung function, cough peak flow, respiratory muscle strength, nasal respiratory pressures, functional capacity, muscle fatigue, cognitive function, as well as surface electromyography of respiratory muscles during active and assisted breathing curves using transcranial magnetic stimulation (TMS), cortical excitability, central tissue oxygenation, respiratory muscle tissue oxygenation, functionality and disease progression, motor control and muscle performance, fatigue and dyspnea, sleep analysis, quality of life, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes; diagnosis of ALS according to the revised El Escorial criteria;
* Age between 18 and 80 years;
* Forced Vital Capacity greater than 50% of predicted;
* Sniff nasal inspiratory pressure greater than 40 cmH2O;
* A telephone number to contact the care team and who signed the study consent form.

Exclusion Criteria:

* Subjects who are unable to understand or perform any of the study procedures;
* Subjects who do not agree to participate or voluntarily request withdrawal from the study at any time;
* Subjects with cardiac, respiratory, or musculoskeletal comorbidities;
* Subjects using invasive mechanical ventilation;
* Subjects with a tracheostomy;
* Subjects with a pacemaker;
* Subjects with metallic brain implants or other electronic implants;
* Subjects with a cochlear implant;
* Subjects with epileptic activity or a history of epilepsy, or a family history of epilepsy;
* Subjects with a history of stroke or tumor;
* Subjects prone to severe hemodynamic fluctuations, acute infectious processes, and/or inflammatory conditions;
* Pregnant women at the time of recruitment;
* Subjects who are unable to complete the intervention protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cortical excitability assessed via TMS | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  Cortical excitability assessed by means of Transcranial Magnetic Stimulation measuring motor evoked potentials, cortical inhibition and duration of the cortical silent period
Cortical tissue oxygenation | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  Assessment of cortical tissue oxygenation using brain coupled near-infrared spectroscopy technique coupled to the brain to monitor cerebral oxygenation and regional cerebral oxygen saturation.
Electromyographic activity of specific respiratory muscles | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed through Electromyography of the sternocleidomastoid, scalene, parasternal, hemidiaphragm and rectus abdominis muscles

SECONDARY OUTCOMES:
Respiratory function assessed by spirometry | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed using spirometry
Maximum Inspiratory and Expiratory Pressure | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed by assessing maximum inspiratory and expiratory pressure, Sniff Nasal Inspiratory Pressure and Sniff Nasal Expiratory Pressure curves
Cough Peak Flow | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed through Cough Peak Flow values
Respiratory muscle oxygenation via near-infrared spectroscopy | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed using the near-infrared spectroscopy technique coupled to the scalene and parasternal muscles
Peripheral upper limb muscle activity assessed via electromyography | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed through a protocol for assessing muscle activity positioned in the Lower Trapezius, Anterior Deltoid, Biceps Brachii (medial head), Triceps Brachii (lateral head), Brachioradialis, Extensor Carpi Radialis Longus, Abductor Pollicis Brevis and Upper Trapezius muscles, bilaterally
Functionality and disease progression | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed using the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised which has 12 items with a score from zero to 4, and its total score can range from zero to 48, where 48 means normal functionality and zero, severe disability
Fatigue Severity | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed using the Fatigue Severity Scale comprises nine statements ranging from 1 to 7, with 7 being the maximum level of agreement with the statement, with a minimum score of 9 and a maximum of 63, with values equal to or greater than 28 indicating fatigue
Dyspnea assessed via Modified Borg Scales | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  The Modified Borg scale is numbered from 0 to 10, with each number referring to a textual description of the degree of respiratory fatigue, with 0 as the minimum and 10 as the maximum respiratory discomfort
Quality of sleep assessment | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed using the Mini-Sleep Questionnaire
Quality of life assessed using the Brief ALS-specific Quality of Life Questionnaire | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed using the Brief Specific Quality of Life Questionnaire for ALS Patients
Subjective assessment of stimulation-related effects | From the date of randomization (1 week before the start of the intervention) up to 6 months (follow-up)
  This outcome will be assessed through a questionnaire about effects such as itching, tingling, redness of the skin, drowsiness, concentration problems, headache, fatigue, dizziness and others, indicating the intensity of these sensations on a scale of 1 to 4 (1 being none, 2 being mild, 3 being moderate and 4 being strong) and whether these effects are related to the stimulation, using a Likert scale from 1 (no relation) to 5 (strongly related)

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (2):
  - Universidade de Brasília - Campus Ceilândia, Brasília, Federal District
  - PneumoCardioVascular Lab - HUOL/UFRN, Natal, Rio Grande do Norte
- Chile (2):
  - Universidad Autónoma de Chile, Santiago, Santiago Metropolitan
  - Universidad do Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided